CLINICAL TRIAL: NCT05366673
Title: Effect of Massage Therapy on Fatigue and Sleep Quality in Patients With Heart Failure in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TYVH109
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2022-08

CONDITIONS: Massage; Heart Failure
Keywords: heart failure; massage; fatigue; sleep quality
MeSH Terms: conditions — Heart Failure; Fatigue; Sleep Initiation and Maintenance Disorders | interventions — Massage

STUDY DESIGN:
Intervention Model Description: Massage
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage therapy (Experimental): Patients will receive massage therapy for 10 minutes, once per day from the first day to the seventh day of admission to the intensive care unit.
  Interventions: Other: massage
- Control group (No Intervention): Patients will maintain usual care.

INTERVENTIONS:
Other: massage — Perform a 10-minute back massage every day for a week
  Arms: Massage therapy

SUMMARY:
The purpose of this study was to explore the effect of massage therapy on fatigue and sleep quality in patients with heart failure in the intensive care unit. The study design was a randomized control trial and repeated measurements. A convenience sampling was used to recruit heart failure patients with New York Heart Association (NYHA) II-III from the intensive care unit of a regional teaching center. In addition to routine turning, patients in the experimental group received daily back massage intervention for 10 minute, once a day; the control group maintained usual care. The data collection included three time points: baseline, 4th and 7th day after the intervention. Research tools include basic personal data, Piper fatigue scale and Pittsburgh sleep quality scale.

DETAILED DESCRIPTION:
The purpose of this study was to explore the effect of massage therapy on fatigue and sleep quality in patients with heart failure in the intensive care unit. The study design was a randomized control trial and repeated measurements. A convenience sampling was used to recruit heart failure patients with New York Heart Association (NYHA) II-III from the intensive care unit of a regional teaching center. In addition to routine turning, patients in the experimental group received daily back massage intervention for 10 minute, once a day; the control group maintained usual care. The data collection included three time points: baseline, 4th and 7th day after the intervention. Research tools include basic personal data, Piper fatigue scale and Pittsburgh sleep quality scale. Data will be analyzed by descriptive statistics, chi-square test, Pearson product correlation, one-way ANOVA, independent sample t test, repeated measure ANOVA, and generalized estimating equation (GEE)。

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure diagnosed by a physician and grade II to III according to NYHA classification, and those who can perform massage therapy after the physician's evaluation
* Over 20 years old
* A person who has a clear consciousness and can communicate
* Those who are willing to accept the implementation of this research plan

Exclusion Criteria:

* People with sleep disorders
* People with mental or cognitive impairment
* Patients who use sedatives or neuroleptics
* Patients with unstable angina, myocardial infarction, and unstable vital signs
* Those who are unconscious and unable to communicate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Changes in Piper Fatigue Scale score | baseline, 4 day, 7 day
  Changes from baseline Piper Fatigue Scale score at 4 days, 7 days. Piper Fatigue Scale contains 15 items. Each item score ranges 0 to 3 with a total score ranged from 0 to 45, higher scores indicate higher fatigue levels.
Changes in Verran and Snyder-Halpern sleep quality scale | baseline, 4 day, 7 day
  Changes from baseline Verran and Snyder-Halpern sleep quality Scale score at 4 days, 7 days. Verran and Snyder-Halpern sleep scale includes 15 items. Each item score ranges from 0-100. Higher score indicates poor sleep.

SECONDARY OUTCOMES:
Changes in Hospital Anxiety and depression scale score | baseline, 4 day, 7 day
  Changes from baseline Hospital Anxiety and depression Scale score at 4 days, 7 days. Hospital Anxiety and Depression Scale includes 14 items, 2 subscales. Each item score ranges from 0 to 3 with a total score of 0-21 for anxiety and depression subscale. Higher score indicates high anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Fu Chiou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- Taipei Veterans General Hospital Taoyuan Branch, Taoyuan District, Taiwan

REFERENCES:
- [Background] Polikandrioti M, Kalafatakis F, Koutelekos I, Kokoularis D. Fatigue in heart failure outpatients: levels, associated factors, and the impact on quality of life. Arch Med Sci Atheroscler Dis. 2019 May 28;4:e103-e112. doi: 10.5114/amsad.2019.85406. eCollection 2019. PMID 31211277
- [Background] Akerstedt T, Hume K, Minors D, Waterhouse J. The subjective meaning of good sleep, an intraindividual approach using the Karolinska Sleep Diary. Percept Mot Skills. 1994 Aug;79(1 Pt 1):287-96. doi: 10.2466/pms.1994.79.1.287. PMID 7991323
- [Background] Klip A, Ramlal T, Bilan PJ, Cartee GD, Gulve EA, Holloszy JO. Recruitment of GLUT-4 glucose transporters by insulin in diabetic rat skeletal muscle. Biochem Biophys Res Commun. 1990 Oct 30;172(2):728-36. doi: 10.1016/0006-291x(90)90735-6. PMID 2241964
- [Background] Backus D, Manella C, Bender A, Sweatman M. Impact of Massage Therapy on Fatigue, Pain, and Spasticity in People with Multiple Sclerosis: a Pilot Study. Int J Ther Massage Bodywork. 2016 Dec 9;9(4):4-13. doi: 10.3822/ijtmb.v9i4.327. eCollection 2016 Dec. PMID 27974947
- [Background] Chen WL, Liu GJ, Yeh SH, Chiang MC, Fu MY, Hsieh YK. Effect of back massage intervention on anxiety, comfort, and physiologic responses in patients with congestive heart failure. J Altern Complement Med. 2013 May;19(5):464-70. doi: 10.1089/acm.2011.0873. Epub 2012 Nov 27. PMID 23186129
- [Background] Chen LX, Ji DH, Zhang F, Li JH, Cui L, Bai CJ, Liu H, Liang Y. Richards-Campbell sleep questionnaire: psychometric properties of Chinese critically ill patients. Nurs Crit Care. 2019 Nov;24(6):362-368. doi: 10.1111/nicc.12357. Epub 2018 Jul 30. PMID 30062842
- [Background] Chen LH, Li CY, Shieh SM, Yin WH, Chiou AF. Predictors of fatigue in patients with heart failure. J Clin Nurs. 2010 Jun;19(11-12):1588-96. doi: 10.1111/j.1365-2702.2010.03218.x. PMID 20579199
- [Background] Conley S, Feder S, Redeker NS. The relationship between pain, fatigue, depression and functional performance in stable heart failure. Heart Lung. 2015 Mar-Apr;44(2):107-12. doi: 10.1016/j.hrtlng.2014.07.008. Epub 2015 Jan 6. PMID 25576085
- [Background] Drouot X, Quentin S. Sleep Neurobiology and Critical Care Illness. Sleep Med Clin. 2016 Mar;11(1):105-13. doi: 10.1016/j.jsmc.2015.10.001. PMID 26972037
- [Background] Evangelista LS, Moser DK, Westlake C, Pike N, Ter-Galstanyan A, Dracup K. Correlates of fatigue in patients with heart failure. Prog Cardiovasc Nurs. 2008 Winter;23(1):12-7. doi: 10.1111/j.1751-7117.2008.07275.x. PMID 18326992
- [Background] Hayhoe B, Kim D, Aylin PP, Majeed FA, Cowie MR, Bottle A. Adherence to guidelines in management of symptoms suggestive of heart failure in primary care. Heart. 2019 May;105(9):678-685. doi: 10.1136/heartjnl-2018-313971. Epub 2018 Dec 4. PMID 30514731
- [Background] Heo S, McSweeney J, Tsai PF, Ounpraseuth S. Differing Effects of Fatigue and Depression on Hospitalizations in Men and Women With Heart Failure. Am J Crit Care. 2016 Nov;25(6):526-534. doi: 10.4037/ajcc2016909. PMID 27802954
- [Background] Huang HW, Zheng BL, Jiang L, Lin ZT, Zhang GB, Shen L, Xi XM. Effect of oral melatonin and wearing earplugs and eye masks on nocturnal sleep in healthy subjects in a simulated intensive care unit environment: which might be a more promising strategy for ICU sleep deprivation? Crit Care. 2015 Mar 19;19(1):124. doi: 10.1186/s13054-015-0842-8. PMID 25887528
- [Background] Fredriksson-Larsson U, Alsen P, Karlson BW, Brink E. Fatigue two months after myocardial infarction and its relationships with other concurrent symptoms, sleep quality and coping strategies. J Clin Nurs. 2015 Aug;24(15-16):2192-200. doi: 10.1111/jocn.12876. Epub 2015 May 19. PMID 25988847
- [Background] Iyngkaran P, Liew D, Neil C, Driscoll A, Marwick TH, Hare DL. Moving From Heart Failure Guidelines to Clinical Practice: Gaps Contributing to Readmissions in Patients With Multiple Comorbidities and Older Age. Clin Med Insights Cardiol. 2018 Dec 4;12:1179546818809358. doi: 10.1177/1179546818809358. eCollection 2018. PMID 30618487
- [Background] Nahmias AJ, Naib ZM, Josey WE, Franklin E, Jenkins R. Prospective studies of the association of genital herpes simplex infection and cervical anaplasia. Cancer Res. 1973 Jun;33(6):1491-7. No abstract available. PMID 4352387
- [Background] Jeon S, Redeker NS. Sleep Disturbance, Daytime Symptoms, and Functional Performance in Patients With Stable Heart Failure: A Mediation Analysis. Nurs Res. 2016 Jul-Aug;65(4):259-67. doi: 10.1097/NNR.0000000000000169. PMID 27362512
- [Background] Sable A, Sivabalan T, Shetti AN. Effectiveness of Back Massage on Sleep Pattern among Patients with Congestive Cardiac Failure. Iran J Nurs Midwifery Res. 2017 Sep-Oct;22(5):359-362. doi: 10.4103/ijnmr.IJNMR_142_16. PMID 29033989